CLINICAL TRIAL: NCT00943943
Title: G-CSF and Plerixafor With Sorafenib for Acute Myelogenous Leukemia With FLT3 Mutations
Brief Title: Granulocyte-colony Stimulating Factor (G-CSF) and Plerixafor Plus Sorafenib for Acute Myelogenous Leukemia (AML) With FLT3 Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry); Genzyme, a Sanofi Company (Industry); Amgen (Industry); National Cancer Institute (NCI) (NIH); Georgia Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0501; R01FD003733 (FDA); R21CA143805 (NIH); NCI-2009-01512 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Acute Myelogenous Leukemia; Leukemia
Keywords: acute myelogenous leukemia; AML; Leukemia; myeloid leukemias; mutated fms-like tyrosine kinase receptor-3; FLT3 Mutations; G-CSF; Granulocyte Colony Stimulating Factor; Filgrastim; Neupogen; Plerixafor; Mobozil; Sorafenib; BAY 43-9006
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Leukemia, Myeloid | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; plerixafor; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- G-CSF and Plerixafor with Sorafenib (Experimental): G-CSF 10 mcg/kg adjusted body weight subcutaneous injection. Plerixafor fixed dose of 240 mcg/kg adjusted body weight subcutaneous injection in abdomen. Patients will receive the 1st doses of G-CSF and Plerixafor on day 1. G-CSF and Plerixafor every other day for 7 total doses, repeated every 28 days. Sorafenib starting dose 400 mg twice daily orally after G-CSF/Plerixafor injections.
  Interventions: Drug: G-CSF; Drug: Plerixafor; Drug: Sorafenib

INTERVENTIONS:
Drug: G-CSF — 10 microgram/kg subcutaneous injection based on adjusted ideal body weight and administered in the evening (prior to the Plerixafor). The 1st dose on day -1 and every other day for 7 total doses. G-CSF administration of 7 every-other-day doses will be repeated every 28 days.
  Other Names: Granulocyte Colony Stimulating Factor; Filgrastim; Neupogen
Drug: Plerixafor — A fixed dose of 240 mcg/kg subcutaneous injection in the abdomen, calculated on ideal body weight. The 1st dose on day -1 and every other day for 7 total doses. Plerixafor administration of 7 every-other-day doses will be repeated every 28 days.
  Other Names: Mobozil
Drug: Sorafenib — First dose will be given right after G-CSF and plerixafor injections. Drug doses will be separated by intervals of approximately 12 hours (+/-2 hours).
  Dose Level 0 = 400 mg orally twice daily.
  Other Names: Nexavar; BAY 43-9006

SUMMARY:
The goal of this clinical research study is to learn the most tolerable dose of Nexavarâ (sorafenib) when given in combination with Mobozilâ (plerixafor) and Neupogenâ (filgrastim) to patients with AML. The safety of this combination will also be studied.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
The Study Drugs:

Sorafenib is a type of drug called a multikinase inhibitor. It is designed to interfere with the parts of cancer cells that are involved in the sending of chemical messages and helping the cells divide and grow, which may block the formation of tumors and cause cell death.

Filgrastim promotes the growth of white blood cells, which help to fight infections.

Plerixafor is designed to help move stem cells from the bone marrow to the blood.

Study Drug Dose Level:

If participant is found to be eligible to take part in this study, they will be assigned to a dose level and schedule of sorafenib based on when they joined this study. Up to 5 dose levels and schedules will be tested. Three (3) participants will be enrolled at each dose level for Phase I of the study. The first group of participants will receive dose level "0" of sorafenib. If unacceptable side effects are seen, a dose lower than level "0" will be tried. If no side effects are seen, the next group of 3 participants will be placed on a higher dose level, called Level "1." Each new group will either receive a higher or lower dose of sorafenib or take it more or less often than the group before it, based on whether intolerable side effects are seen. This will continue until the best tolerable dose and schedule of sorafenib is found. Once the best tolerable dose and/or schedule is found, the last 10 participants will be enrolled and will take sorafenib at that dose and schedule. This last group of 10 is considered the early Phase II part of the study.

Each group will receive the same dose level and schedule of filgrastim and plerixafor.

Study Drug Administration:

Participant will receive filgrastim and plerixafor by injection through a needle under the skin on Day 1 (the day the study starts) and then every other day for a total of 7 doses. The injections will be given in the morning. After day one, the injections may be done at participant's home. Participant's study doctor will meet with them one-on-one to discuss how the drug will be given.

On Day 1, participant will begin taking their dose of sorafenib by mouth every other day, once a day, or twice a day, depending on when they join the study.

* If participant is taking sorafenib every other day, during Cycle 1 they will start taking it 12 hours after the filgrastim and plerixafor injections (the next morning) .
* If participant is taking sorafenib every day, they will take it at the same time every morning. The first time participant takes sorafenib during Cycle 1 will be 12 hours after the first filgrastim and plerixafor injections.
* If participant is taking sorafenib twice a day, during Cycle 1 they will start taking it 12 hours after the filgrastim and plerixafor injections and then every 12 hours.

Participant will take sorafenib without food, at least 1 hour before or 2 hours after eating. If participant misses a dose, they should not take double the dose next time to make up for the missed dose.

These 28 days are one "study cycle".

Participant is allowed to take hydroxyurea or other treatments to control high white blood cell counts.

Study Drug Diary:

Participant will be given a study drug diary that they will be expected to fill out whenever they take study drugs at home. A staff member will explain to participant how to fill out the diary. The study staff will review the diary with participant at every study visit and they will be given a new diary at the beginning of every cycle they start.

Study Visits:

Every week for the first 6 weeks and then every 4-8 weeks until participant leaves the study, the following tests and procedures will be performed:

* Participant will have a physical exam, including measurement of their weight, and vital signs.
* Participant will have a bone marrow aspiration and biopsy done before treatment starts and once somewhere between day 14 and day 17 after the first Sorafenib administration. Another bone marrow sample will be collected between days 24 and 28.
* If participant continues on study, another bone marrow sample will be collected after the third cycle.
* Blood (about 1 teaspoon) will be drawn every 2-4 days for routine tests while participant is taking the study drugs and once a week on days they are not taking the study drugs Plerixafor and Neupogen.
* During the first week, blood (about 1 teaspoon) will be drawn to check the status of the disease before each dose of the filgrastim and plerixafor combination and again 4 to 8 hours after receiving the study drugs. If participant's doctor feels it is needed, additional blood may be drawn after the 2nd blood draw to check the status of the disease. If participant's doctor feels it is needed, these blood draws may continue after the first week if the disease is not responding.

Length of Study:

Participant may continue taking the study drugs for up to 6 cycles (about 6 months). If participant is in complete remission, partial remission, or complete remission with incomplete platelet count recovery after 6 months with no intolerable side effects, their doctor may discuss continuing on the study with them. Participant will be taken off study if the disease gets worse or intolerable side effects occur.

Follow-up Visits:

If participant is in complete remission, and if their doctor thinks it is in their best interest, they may have follow-up visits about every 3 months until the study closes.

* Blood (about 2 teaspoons) will be drawn for routine tests.
* Participant will have a bone marrow biopsy and/or aspirate to check the status of the disease.

End-of-Study Visit:

Participant will have an end-of-study visit about 30 days after their last dose of the study drugs. At this visit, the following tests and procedures will be performed:

* Participant will have a physical exam, including measurement of their weight and vital signs.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* Participant will have a bone marrow aspirate and biopsy to check the status of the disease.

This is an investigational study. Sorafenib is FDA-approved and commercially available for treatment of advanced renal cell cancer (RCC) and hepatocellular cancer (HCC) that cannot be removed by surgery. Its use in patients with AML is investigational.

Plerixafor is FDA-approved and commercially available for use in boosting the number of hematopoietic stem cells (HSC) for stem cell collection and transplants (in combination with filgrastim) in participants with non-Hodgkin's lymphoma (NHL) and multiple myeloma (MM). Its use in participants with AML is investigational.

Filgrastim (NeupogenÒ) is FDA-approved and commercially available for use in boosting white blood cell production in participants with low blood cell counts caused by chemotherapy (nonmyeloid malignancies, acute myeloid leukemia, and bone marrow transplantation), treating severe chronic neutropenia (SCN-low blood counts), and boosting production of hematopoietic progenitor cells in patients undergoing peripheral blood progenitor cell (PBPC) collection.

Up to 28 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be 18 years of age or older.
2. Patients must have relapsed/refractory leukemia with FLT3 (ITD) mutations. Patients with AML FLT3 mutations who are not eligible for frontline standard therapy, or who refuse to be treated with intensive chemotherapy, may be eligible.
3. Serum biochemical values with the following limits unless considered due to leukemia: creatinine </= 1.5 mg/dl; total bilirubin </= 1.5 mg/dL, unless increase is due to hemolysis or congenital disorder; or transaminases (SGPT) </= 2.5 x upper limit of normal (ULN)
4. Able to take oral medication.
5. Able to understand and provide signed informed consent.
6. Ejection fraction at screening must be >/=50%.
7. Performance status < 3, unless directly related to leukemic disease process as determined by the Principal Investigator.

Exclusion Criteria:

1. Subjects with acute promyelocytic leukemia.
2. Patients with absolute blast count > 20 k/uL.
3. Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, intrauterine device (IUD), diaphragm, abstinence, or condoms by their partner) over the entire course of the study.
4. Men not willing to maintain adequate contraception with their partner over the entire course of the study.
5. Hypertension > 140 mmHg systolic OR > 90 mmHg diastolic with or without antihypertensive therapy.
6. Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
7. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy. Sorafenib is contraindicated in patients with known severe hypersensitivity to sorafenib or any of the excipients.
8. Known human immunodeficiency virus (HIV) infection or active Hepatitis B or C.
9. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
10. Pulmonary hemorrhage/bleeding event >/= CTCAE Grade 2 within 4 weeks of first dose of study drug.
11. Any other hemorrhage/bleeding event >/= CTCAE Grade 3 within 4 weeks of first dose of study drug.
12. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
13. Currently using St. John's Wort or rifampin.
14. Known or suspected allergy to sorafenib or any agent given in the course of this trial.
15. Active clinically serious and uncontrolled infection > CTCAE Grade 2.
16. Serious non-healing wound, ulcer, or bone fracture.
17. Patients currently receiving any other standard or investigational treatment for their hematologic malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-10-29 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Sorafenib | Participant toxicity rates evaluated at 8 weeks of treatment (2 cycles)
  MTD dose level of Sorafenib where less than two participants (2/3) experience Dose limiting toxicity (DLT), based on Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, is defined as ± Grade 3 nonhematological toxicity or nausea/vomiting (in the absence of appropriate antiemetics) that cannot be explained by intercurrent conditions such as infections and at least possibly related to the combination of agents in study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Andreeff, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org